CLINICAL TRIAL: NCT05472519
Title: Immunopathology of Loeys-Dietz Syndrome
Acronym: I-LoDiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0016
Record Dates: First submitted 2022-06-30; First posted 2022-07-25 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Loeys-Dietz Syndrome
Keywords: Loeys-Dietz Syndrome; immunology; T-Lymphocytes
MeSH Terms: conditions — Loeys-Dietz Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loeys-Dietz syndrome (Other): Patients aged ≥ 5 years with Loeys-Dietz syndrome with a diagnosis confirmed by the presence of a TGF-βR 1 or R2 mutation.
  Interventions: Biological: blood samples
- Healthy Group (Other): Subjects aged ≥ 5 years.
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — Only one visit for each participant: A large majority of visits will be part of patients' usual care.
  * Medical examination : weight, gender, blood pressure, medical history
  * Blood samples : 1 EDTA tube (3 mL) for CBC, 3 heparin tubes (3 × 7 mL) for frozen PBMC, 1 EDTA tube (3 mL) for frozen plasma
Biological: blood samples — Only one visit for each participant:
  * Medical examination : weight, gender, blood pressure, medical history
  * Blood samples : 1 EDTA tube (3 mL) for CBC, 3 heparin tubes (3 × 7 mL) for frozen PBMC, 1 EDTA tube (3 mL) for frozen plasma

SUMMARY:
Loeys-Dietz syndrome (LDS) is a rare vascular genetic disorder (estimated prevalence 1/25,000-1/100,000) due primarily to mutations in the Transforming growth factor beta (TGF-β) cytokine receptor 1 and 2 genes. In addition to a common vascular phenotype with Marfan syndrome (dilatation of the ascending aorta, arachnodactyly, lens dislocation), patients present specific malformations (bifid uvula, hypertelorism, tortuous arteries) and immuno-allergic manifestations (asthma, eczema, food allergy, eosinophilic esophagitis, chronic inflammatory bowel disease).

Pathophysiologically, LDS appears to be associated with hyperactivation of the intracellular TGF-β signaling pathway in a manner similar to Marfan syndrome, as evidenced by increased intracellular phosphorylated Smad2/3 (pSmad2/3) in lymphocytes. The immuno-allergic complications appear paradoxical because of the major immunosuppressive role of this cytokine on lymphoid and myeloid immune lineages.

The biological description of immunological abnormalities associated with LDS is based on a single 2013 study that found increased regulatory T (Treg) and Th2 lymphocyte polarizations, as well as increased circulating eosinophil and total IgE levels.

In order to better understand the underlying mechanisms, the investigators propose to perform a descriptive clinical-biological study to identify and study the immune subpopulations most impacted by the causative mutations of LDS.

ELIGIBILITY:
Inclusion Criteria:

For patients with Loeys-Dietz syndrome:

* Patients aged ≥ 5 years with Loeys-Dietz syndrome with a diagnosis confirmed by the presence of a TGF-βR 1 or R2 mutation known to be pathogenic to patients.
* Free, informed and signed consent from the patient or both parents or legal guardians for minor patients.
* Patient affiliated to a social security system or similar.

For healthy volunteers:

* Subjects aged ≥ 5 years.
* Free, informed and signed consent of the witness, or if applicable of both parents or legal representatives for minors.
* Patient affiliated to a social security system or similar.

Exclusion Criteria:

For patients with Loeys-Dietz syndrome:

* Patient with an evolving or recently healed (< 3 months) cancer that could alter the immunologic profile.
* Patient with an evolving or recently healed (< 3 months) infection that could alter the immunologic profile.
* Patient with a weight of less than 20 kg.
* Pregnant woman.
* Patient participating in another research study with an exclusion period exclusion period still in progress.

For healthy volunteers:

* Subject with an active or recently cured (< 3 months) cancer that could alter the immunologic profile.
* Subject with an active or recently healed (< 3 months) infection that could alter the immunological profile.
* Patient with a weight of less than 20 kg.
* Pregnant woman.
* Subject participating in another research study with an exclusion period exclusion period still in progress.
* Persons under court protection.

Ages: 5 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Percentage of circulating TFH lymphocyte subpopulation. | Day 1
  Measured from the Blood samples of each patients / volunteers.

SECONDARY OUTCOMES:
Intracellular pSmad2/3 labeling level of circulating TFH lymphocytes. | Day 1
  Measured from the Blood samples of each patients / volunteers.
Identification of Immuno-allergic pathologies | Day 1
  Identification of Immuno-allergic, serious infectious pathologies (diagnostic criteria, severity criteria, treatment, current activity) in LDS patients.
Identification of serious infectious pathologies | Day 1
  Identification of serious infectious pathologies (diagnostic criteria, severity criteria, treatment, current activity) in LDS patients.
Identification of Vascular complications | Day 1
  Identification of Vascular, morpho-skeletal complications (diagnostic criteria, severity criteria, treatment, current activity) current course) in patients with LDS.
Identification morpho-skeletal complications | Day 1
  Identification of morpho-skeletal complications (diagnostic criteria, severity criteria, treatment, current activity) current course) in patients with LDS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant / Centre de Compétences pour le syndrome de Marfan et apparentés, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided